CLINICAL TRIAL: NCT05612009
Title: Assessment of Different Imaging Systems for Dental Plaque Scoring: an In-vivo Study
Brief Title: Assessment of Different Imaging Systems for Dental Plaque Scoring
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: S1s7s9s3
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Dental Plaque Imaging Methods
Keywords: dental plaque; dental photography; digital scanning system; fluorecam; Turesky Modified Quigley Hein Plaque Index
MeSH Terms: conditions — Dental Plaque | interventions — Toothpastes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — dental plaque samples of volunteers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- 1. Signal Expert Protection: After scoring clinically and with dental plaque imaging methods, Signal Expert Protection toothpaste was given to 10 volunteers.
  Interventions: Combination Product: Toothpastes
- 2. Colgate Hemp Seed Oil: After scoring clinically and with dental plaque imaging methods, Colgate Hemp Seed Oil toothpaste was given to 10 volunteers.
  Interventions: Combination Product: Toothpastes
- 3. Gumgumix: After scoring clinically and with dental plaque imaging methods, Gumgumix toothpaste was given to 10 volunteers.
  Interventions: Combination Product: Toothpastes

INTERVENTIONS:
Combination Product: Toothpastes — Signal Expert Protection: Conventional toothpaste including Sodium Lauryl Sulphate and fluoride.
  Colgate Hemp Seed Oil: Herbal toothpaste including hemp seed oil and also fluoride.
  Gumgumix: Herbal toothpaste including ginger extract (no fluoride).
  Other Names: Signal Expert Protection, Colgate Hemp Seed Oil, Gumgumix

SUMMARY:
The aim of this study was to analyze the correlation between the dental plaque indices measured different imaging systems and conventional clinical indices that assess dental plaque. From among the patients who visited Marmara University, Faculty of Dentistry 30 adults between the age of 18-30, who had under 3 DMFT scores, were selected for full-mouth imaging. Digital dental photography, digital scanning system and fluorecam methods were used for taking intraoral images. The Turesky Modified Quigley Hein Plaque Index (TMQHPI) was scored both by the clinical examination method and on the images taken. The correlations between the clinical examinaton, digital photography, digital scanning system and fluorecam scores were analyzed. Maxillary and mandibulary anterior teeth's buccal surfaces were scored to TMQHPI after using disclosing agent.

DETAILED DESCRIPTION:
The study was performed with 30 adult patients aged between 18-35, recruited from among the outpatients who visited the Marmara University, Faculty of Dentistry, Restorative Dentistry Department, agreed to the terms of the experiment, had a DMFT score 3 or lower, and had relatively even teeth arrangement. Among patients, those with orthodontic bracket placed, severe crowding of teeth not visually verified in the photograph, fixed or implant restoration installed, more than 3 DMFT score, and serious systemic diseases were excluded from the study.

In order to standardize the study, the volunteers were informed that they shouldn't eat any nutrients and do oral hygiene practices after dinner. Visualization of plaque samples formed in the mouth at least 8-12 hours between 08:30 and 10:00 a.m. in the morning and collecting dental plaque samples for microbiological examination were performed after the volunteers signed the informed consent form. The Turesky Modified Quigley Hein Plaque Index (TMQHPI) was scored both by the clinical examination method and on the images taken. The correlations between the manuel examinaton, digital photography, digital scanning system and fluorecam scores were analyzed. Maxillary and mandibulary anterior teeth's buccal surfaces were scored to TMQHPI after using disclosing agent. Using the standard toothbrush provided to the volunteers, they were asked to brush their teeth twice a day for 21 days with the recommended brushing method. After 21 days, dental plaque scoring and imaging procedure was repeated and dental plaque samples were collected again and placed in Eppendorf tubes. Eppendorf tubes were kept at -80 °C during the study. Bacterial changes in the samples taken on Day 0 and Day 21 were examined by Polymerase Chain Reaction (PCR) method in Marmara University Faculty of Medicine, Department of Clinical Microbiology. The levels in plaque samples of Streptococcus mutans, Lactobacillus acidophilus, Actinomyces viscosus, , Candida albicans, Staphylococcus aerus, were measured.

ELIGIBILITY:
Inclusion Criteria:

The volunteers between the ages of 18-35, No systemic disease, Teeth that do not contain hereditary, morphological, drug-induced structural changes, Not using orthodontic wires and appliances, Having a DMFT score of 3 and less than 3, Have not received antibiotic treatment in the last 6 weeks, Not using mouthwash in the last 6 weeks, Without dental calculus, Oral hygiene habits are similar to each other, University student or graduate, Thirty volunteers who were conscious of being able to understand and apply the guidelines set forth in the study were included.

Exclusion criteria:

Among volunteers, those with orthodontic bracket placed, severe crowding of teeth not visually verified in the photograph, fixed or implant restoration installed, more than 3 DMFT score, and serious systemic diseases were excluded from the study.

Ages: 18 Years to 35 Years | Sex: All
Age Groups: Adult
Study Population: The study was performed with 30 adult male and female patients aged between 18-35, recruited from among the outpatients who visited the Marmara University, Faculty of Dentistry, Restorative Dentistry Department, agreed to the terms of the experiment, had a DMFT score 3 or lower, and had relatively even teeth arrangement. Among patients, those with orthodontic bracket placed, severe crowding of teeth not visually verified in the photograph, fixed or implant restoration installed, more than 3 DMFT score, and serious systemic diseases were excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
1. Dental plaque scoring clinically before staining agent | 15 minutes
  Dental plaque of the volunteer's anterior teeth were scored to Turesky Modified Quigley Hein Plaque Index
2. Dental plaque scoring clinically after applying staining agent | 15 minutes
  Dental plaque of the volunteer's anterior teeth were scored to Turesky Modified Quigley Hein Plaque Index
3.Dental plaque scoring after applying staining agent on the taken images with FluoreCam | 45 minutes
  Dental plaque of the volunteer's anterior teeth were scored on the images taken with FluoreCam to Turesky Modified Quigley Hein Plaque Index
4. Dental plaque scoring after applying staining agent on the taken images with Digital Camera | 45 minutes
  Dental plaque of the volunteer's anterior teeth were scored on the images taken with FluoreCam to Turesky Modified Quigley Hein Plaque Index
5. Dental plaque scoring after applying staining agent on the taken images with Intraoral Scanner | 1 hour
  Dental plaque of the volunteer's anterior teeth were scored on the images taken with Intraoral Scanner to Turesky Modified Quigley Hein Plaque Index

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Department of Restorative Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after the publication of the article.
Supporting Information: Study Protocol, ICF
Time Frame: data will be available in 2 years.
Access Criteria: all researchers may access the data of this study